CLINICAL TRIAL: NCT03803644
Title: A Phase 1, Two-part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Dosing of CC-92480 and to Explore the Effect of Food on the Bioavailability of CC-92480 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of Single Ascending Doses of CC-92480 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-92480-CP-001; U1111-1224-6768 (Registry Identifier: WHO)
Record Dates: First submitted 2018-12-17; First posted 2019-01-14 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteer
Keywords: Healthy Subjects; CC-92480; Food Effect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Administration of CC-92480 - Part 1 (Experimental): dose escalation
  Interventions: Drug: CC-92480
- Administration of CC-92480 under fasted conditions - Part 2 (Experimental): Food effect
  Interventions: Drug: CC-92480
- Administration of CC-92480 under fed conditions - Part 2 (Experimental): food effect
  Interventions: Drug: CC-92480

INTERVENTIONS:
Drug: CC-92480 — Part 1 dose escalation
  Arms: Administration of CC-92480 - Part 1
Drug: CC-92480 — CC-92480
  Arms: Administration of CC-92480 under fasted conditions - Part 2; Administration of CC-92480 under fed conditions - Part 2

SUMMARY:
This is a two-part study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of CC-92480 and explore the effect of food on the bioavailability of CC-92480 in healthy subjects.

Part 1:

Part 1 is a single-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, and pharmacodynamics (PD) of CC-92480 following administration of single oral doses in healthy adult subjects. Part 1 will consist of escalating single doses in sequential groups. Approximately 40 subjects will be enrolled into 5 planned dose level cohorts. Each dose level cohort will consist of 8 subjects; 6 subjects will receive CC-92480 and 2 subjects will receive placebo according to the randomization schedule.

Part 2 Part 2 is a single-center, open-label, randomized, 2-period, 2-way crossover study to explore the effect of food (Food and Drug Administration [FDA] standard high-fat breakfast) on the single-dose PK of CC-92480 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Must understand and voluntarily sign a written informed consent form (ICF) prior to any study-related assessments/procedures being performed.
2. Must be able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
3. Be a healthy male or female of non-childbearing potential of any race, between 18 to 55 years of age (inclusive) at the time of signing the ICF, and in good health as determined by the screening history and PE.
4. Agrees to abide by the requirements and restrictions outlined in the CC-92480 Pregnancy Prevention Plan for Subjects in Clinical Trials.
5. For males: Agree to use barrier contraception not made of natural (animal) membrane (eg, latex or polyurethane condoms are acceptable) when engaging in sexual activity with a female of childbearing potential (FCBP) 1 while on study medication, and for at least 3 months after the last dose of study medication. For females: Female subjects must have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 months without menses before screening, with a plasma follicle-stimulation hormone [FSH] level of > 40 IU/L at screening).
6. Must have a body mass index between 18 and 33 kg/m2 (inclusive) at the time of signing the ICF.
7. No clinically significant laboratory test results as determined by the investigator.
8. At the screening visit, must be afebrile, with supine systolic BP: 90 to 140 mmHg, supine diastolic BP: 50 to 90 mmHg, and pulse rate: 40 to 90 bpm. Eligibility criteria for vital signs performed during check-in and/or predose on Day 1 will be at the discretion of the Investigator. Repeat vital signs may be measured at Investigator discretion.
9. Must have a normal or clinically-acceptable 12-lead ECG at screening. Male subjects must have a corrected QT interval using Fridericia's formula (QTcF) value ≤ 430 msec. Female subjects must have a QTcF value ≤ 450 msec.
10. Subject must agree and be willing to consume a standard high-fat meal (which may contain gluten), for Part 2 subjects only.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. History of any clinically significant and relevant neurological, GI, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders as determined by the Investigator.
2. Any condition that places the subject at unacceptable risk if he or she were to participate in the study, or confounds the ability to interpret data from the study.
3. Use of any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days of the first dose administration.
4. Use of any nonprescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration.
5. Use of CYP3A inducers and inhibitors (including St. John's Wort) within 30 days of the first dose administration.
6. Has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME), eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable. Prior procedures of unclear ADME significance should be reviewed with the Sponsor's Medical Monitor.
7. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
8. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or positive drug screening test reflecting consumption of illicit drugs.
9. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or positive alcohol screen.
10. Known to have serum hepatitis; known to be a carrier of the hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti-HBs), hepatitis B core antibody (anti-HBc), or hepatitis C antibody (HCV Ab); have a positive result to the test for hepatitis B or hepatitis C virus at screening or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening. Subjects whose results are compatible with prior immunization against hepatitis B may be included at the discretion of the Investigator.
11. Exposure to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
12. Use of tobacco- or nicotine-containing products within 3 months prior to Day -1 (Period 1 for Part 2).
13. Vaccination within 30 days of dosing or plans to receive vaccination within 30 days after dosing.
14. Systemic infection within 30 days of dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics- Cmax Part 1 | Day 1
  Maximum plasma concentration of drug
Pharmacokinetics- Tmax Part 1 | Day 1
  Time to maximum plasma concentration
Pharmacokinetics- AUC0-∞ Part 1 | Up to 72 hours after dose administration
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics- AUC0-t Part 1 | Up to 72 hours after dose administration
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration
Pharmacokinetics- AUC0-24 Part 1 | Up to 24 hours after dose administration
  Area under the plasma concentration-time curve from time zero to 24 hours postdose
Pharmacokinetics- AUC-t½ Part 1 | Up to 72 hours after dose administration
  Terminal half-life
Pharmacokinetics- CL/F Part 1 | Up to 72 hours after dose administration
  Apparent total plasma clearance
Pharmacokinetics- Vz/F Part 1 | Up to 72 hours after dose administration
  Apparent total volume of distribution
Pharmacokinetics- Cmax Part 2 | Day 1
  Maximum plasma concentration of drug
Pharmacokinetics- Tmax Part 2 | Day 1
  Time to maximum plasma concentration
Pharmacokinetics- AUC0-∞ Part 2 | Up to 72 hours after dose administration
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics- AUC0-t Part 2 | Up to 72 hours after dose administration
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration
Pharmacokinetics- AUC0-24 Part 2 | Up to 24 hours after dose administration
  Area under the plasma concentration-time curve from time zero to 24 hours post dose
Pharmacokinetics- AUC-t½ Part 2 | Up to 72 hours after dose administration
  Terminal half-life

SECONDARY OUTCOMES:
Adverse Event(s) | From enrollment until at least 28 days after completion of study treatment
  Number of participants with adverse events
Effect of CC-92480 on ECG parameters- Part 1 | Up to day 2
  12-lead ECGs extracted from continuous (Holter) recordings will be used to assess effect of CC-92480 on Qt/QTc ECG parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene
Locations (1):
- Covance-Daytona Beach, Daytona Beach, Florida, United States

REFERENCES:
- [Derived] Wu F, Liu L, Gaudy A, Wang X, Carayannopoulos L, Pourdehnad M, Lamba M. Model based assessment of food and acid reducing agent effects on oral absorption of mezigdomide (CC-92480), a novel cereblon E3 ligase modulator. CPT Pharmacometrics Syst Pharmacol. 2023 Oct;12(10):1473-1484. doi: 10.1002/psp4.13024. Epub 2023 Sep 13. PMID 37705327